CLINICAL TRIAL: NCT06469528
Title: ESCALATion of Medical Therapy Following Multimodality Plaque Evaluation in High-risk Chronic Coronary Syndromes
Acronym: ESCALATE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCH23-187
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
Keywords: Chronic coronary syndromes
MeSH Terms: conditions — Coronary Artery Disease | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Single centre, open-label prospective, randomised controlled trial; patients randomised 1:1 to low-dose colchicine 0.5mg OD vs guideline directed medical therapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose colchicine 0.5mg OD (Experimental): Low dose colchicine 0.5mg OD for 6 months
  Interventions: Drug: Colchicine 0.5 MG
- Guideline directed therapy (No Intervention): Guideline directed therapy; participants will be maintained on maximal tolerated dose of established statin therapy (>4 weeks)

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Low dose daily colchicine
  Arms: Low dose colchicine 0.5mg OD

SUMMARY:
ESCALATE will provide a thorough investigation of how anti-inflammatory therapy, with low-dose colchicine, affects patients with stable coronary artery disease. Using traditional clinical risk factors and multimodality intracoronary imaging, the investigators will identify patients with the greatest clinical risk.

Participants will undergo repeat multimodality intracoronary imaging assessment at 6 months to measure the impact once-daily low-dose colchicine therapy on the structure and function of coronary arteries.

This study will provide valuable insights into how anti-inflammatory therapies, such as colchicine, may improve outcomes in patients with coronary artery disease.

DETAILED DESCRIPTION:
1. Background and study aims

   Despite recent advances, coronary artery disease (CAD) remains the main cause of death worldwide. CAD occurs when the arteries bringing blood to the heart become narrowed by a build-up of fatty material within their walls. If this occurs gradually, it can cause chest discomfort i.e., angina. In a heart attack, the artery wall becomes inflamed and splits causing blood clot formation and an abrupt blockage of flow, resulting in severe pain and damaged heart muscle.

   Current treatments focus on reducing cholesterol, slowing the build-up of fatty material, and rapidly restoring blood flow during a heart attack. Chronic inflammation, acting in tandem with other risk factors, has been identified as playing a central role in CAD progression and its acute manifestations.

   Colchicine is a safe, well-tolerated, anti-inflammatory therapy used in the treatment of gout and other inflammatory conditions. Daily treatment with low-dose colchicine has proven effective in reducing rates of heart attack and death in large clinical trials, but use in routine practice remains low. A contributing factor to this reticence is uncertainty regarding the mechanism through which colchicine provides benefit. This study is designed to address this knowledge gap.
2. Who can participate?

   Patients aged 18 to 90 years old with coronary artery disease and high clinical risk
3. What does the study involve?

Using traditional markers of clinical risk and state-of-the-art imaging from inside the coronary artery, the researchers will identify patients with CAD and the greatest clinical risk. Eligible patients, already established on statin therapy will be allocated to a six-month course of low-dose colchicine plus usual care, or usual care only. Researchers, participants, and usual clinicians will be aware of the allocation during the study.

After 6 months, the researchers will assess the impact of colchicine on the appearance of individual coronary artery lesions, blood flow in the large and small blood vessels of the heart. This study will provide a detailed assessment of colchicine and its mechanism of action in CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent
2. Age 18 to 90 years old
3. Male, or female of non-child-bearing potential
4. Elevated clinical risk, as evidenced by ≥1 of:

   * Previous spontaneous acute myocardial infarction (diagnosed according to the universal MI criteria) with or without persistent ST-segment elevation
   * Previous stroke or intervention for peripheral arterial disease (i.e., evidence of atherosclerotic disease affecting >1 vascular bed)
   * Established diagnosis of diabetes mellitus
   * Systemic Coronary Risk Estimation 2 (SCORE2) or Systemic Coronary Risk Estimation 2 - Older Persons (SCORE2-OP) algorithm 10-year risk of fatal and non-fatal myocardial infarction or stroke >10%
5. Documented evidence of coronary artery disease, with an angiographically moderate stenosis on invasive coronary angiography (30-80%)

   - At least one non-flow limiting (FFR >0.80) moderate lesion with TCFA (minimum fibrous cap thickness of less than or equal to120µm and lipid arc >90°)
6. History of prescribed statin therapy, at a stable dose, for >4 weeks
7. Evidence of residual inflammation at baseline (i.e., high-sensitivity CRP ≥2)

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or of child-bearing potential
2. Symptoms of unstable angina, characterised as: angina at rest; new onset of severe exertional angina (CCS grade III or higher for <4 weeks); or distinct, sudden, intensification of previously stable angina
3. Previous spontaneous acute myocardial infarction (diagnosed according to the universal MI criteria) with or without persistent ST-segment elevation <4 weeks from recruitment
4. Previous coronary artery bypass grafting
5. Known chronic total occlusion of coronary artery
6. Chronic kidney disease with eGFR <50 mL/min/1.73 m2 per MDRD formula or renal replacement therapy at baseline assessment
7. Known active or recurrent hepatic disorder (including cirrhosis, hepatitis B and hepatitis C, or confirmed ALT/AST levels > 3 times ULN or total bilirubin > 2 times ULN) at baseline assessment
8. Symptoms of severe heart failure (systolic or diastolic) with New York Heart Association (NYHA) Functional Classification 3 or 4
9. Moderate or severe valvular heart disease considered likely to require intervention
10. History of blood dyscrasia including anaemia, thrombocytopenia, neutrophilia, leukopenia or other abnormality of blood count at baseline
11. Peripheral neuritis, myositis or marked myo-sensitivity to statins
12. A history of alcohol and/or substance abuse that could interfere with the conduct of the trial
13. Patients with suspected or proven immunocompromised state, including:

    1. those with evidence of Human Immunodeficiency Virus (HIV) infection; Patients on anti-retroviral therapy are excluded
    2. those with any other medical condition which in the opinion of the investigator places the patient at unacceptable risk for participation in immunomodulatory therapy
14. History of hypersensitivity to the study drug or its constituents
15. Patients who have received an investigational drug or device within 30 days (inclusive) of baseline assessment, or who are expected to participate in any other investigational drug or device study during the conduct of this trial
16. Any biologic drugs targeting the immune system (for example, TNF blockers, anakinra, rituximab, abatacept, tocilizumab)
17. Established long-term pharmacotherapy with a strong CYP3A4 inhibitor or a P-glycoprotein inhibitor (P-gpi) (e.g., macrolide antibiotics, ciclosporin, ketoconazole, itraconazole, voriconazole, HIV protease inhibitors, verapamil, diltiazem and disulfiram)
18. Contraindications to intravenous adenosine will exclude patients from adenosine induced hyperaemia
19. Any life-threatening condition with life expectancy <6 months that might prevent the patient from completing the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-24 (Estimated); Primary Completion 2025-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Absolute change in minimal fibrous cap thickness | 6months
  The absolute change (µm) in minimal fibrous cap thickness, in a defined arterial region of interest, as assessed by OCT

SECONDARY OUTCOMES:
Major adverse clinical events | 6 months
  Major adverse cardiovascular event (MACE): Composite of cardiovascular death, non-fatal MI, unplanned revascularisation and ischaemic stroke
Acute kidney injury | 6 months
  AKI secondary to contrast induced nephropathy
Major bleeding events (BARC 3-5) | 6 months
  Periprocedural major bleeding events (BARC 3-5)
Hospitalisation with serious infection | 6 months
  Hospitalisation requiring intravenous antibiotics
% change in minimal fibrous cap thickness | 6 months
  Percentage change in minimal fibrous cap thickness, as determined by OCT, in a defined arterial region of interest
% change in maximal lipid arc | 6 months
  Percentage change in lipid arc, as determined by OCT, in a defined arterial region of interest
Percentage change in lipid index | 6 months
  Percentage change in lipid index, as determined by OCT, in a defined arterial region of interest
Absolute change in maximum lipid core burden index in a 4-mm segment (maxLCBI4mm) | 6 months
  Absolute change in maximum lipid core burden index in a 4-mm segment (maxLCBI4mm), as determined by NIRS, in a defined arterial region of interest
Relative change (%) in maximum lipid core burden index in a 4-mm segment (maxLCBI4mm) | 6 months
  Relative change (%) in maximum lipid core burden index in a 4-mm segment (maxLCBI4mm), as determined by NIRS, in a defined arterial region of interest
Change in total atheroma volume | 6 months
  Change in percent atheroma volume, as determined by IVUS, in a defined arterial region of interest
Absolute and percentage change in coronary flow reserve (CFR) | 6 months
  Absolute and percentage change in coronary flow reserve (CFR), measured in artery of interest
Absolute and percentage change in index of microvascular resistance (IMR) | 6 months
  Absolute and percentage change in index of microvascular resistance (IMR), measured in artery of interest
Absolute and percentage change in vessel fractional flow reserve (FFR) | 6 months
  Absolute and percentage change in vessel fractional flow reserve (FFR), measured in artery of interest
Percentage change in high-sensitivity c-reactive protein (hs-CRP) | 6 months
  Percentage change in high-sensitivity c-reactive protein (hs-CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Pareek, MA MBBS PhD, Principal Investigator — King's College Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No